CLINICAL TRIAL: NCT06045286
Title: High- and Low-dose Radiotherapy Combined With PD-1 Inhibitors for Microsatellite Stable (MSS) Colorectal Liver Metastases (CRLM)
Brief Title: High- and Low-dose Radiotherapy Combined With PD-1 Inhibitors for MSS CRLM
Acronym: HaRyPOT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Lijun Wang, Associate Professor, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HaRyPOT
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Liver Metastases
Keywords: microsatellite stable; PD-1 Inhibitors; abscopal effects
MeSH Terms: interventions — Radiotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High- and Low-dose radiotherapy combined with immunotherapy. (Experimental): All eligible patients will receive high-dose radiotherapy, followed by low-dose radiotherapy combined with PD-1 inhibitor therapy starting within 7 days after completion. The single dose of high-dose radiotherapy will be 6-8 Gy for 3-7 consecutive exposures, and the single dose of low-dose radiotherapy will be 0.5-1.4 Gy for 3-7 consecutive exposures.The PD-1 inhibitor (Zimberelimab) will be administered at the dose recommended in the specification every 3 weeks until disease progression, unacceptable toxicity, and withdrawal of informed consent by the patient.
  Interventions: Radiation: Radiation: High- and Low-dose radiotherapy; Drug: PD-1 Inhibitors

INTERVENTIONS:
Radiation: Radiation: High- and Low-dose radiotherapy — High-dose radiotherapy (6-8Gy×3-7F) followed by low-dose radiotherapy (0.5-1.4Gy×3-7F) starting within 7 days after completion.
Drug: PD-1 Inhibitors — Immunotherapy (Zimberelimab) is given every three weeks within one week after the end of high-dose radiotherapy.

SUMMARY:
This pilot phase I trial aims to investigate the efficacy and safety of high- and low-dose radiotherapy combined with programmed cell death-1 (PD-1) inhibitors in microsatellite stable (MSS) metastatic colorectal cancer (mCRC) that have failed second-line immunotherapy or above.

DETAILED DESCRIPTION:
This pilot phase I trial aims to investigate the efficacy and safety of high- and low-dose radiotherapy combined with programmed cell death-1 (PD-1) inhibitors in microsatellite stable (MSS) metastatic colorectal cancer (mCRC) that have failed second-line immunotherapy or above. 30 participants will be enrolled in this study. All will take part at Jiangsu Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with microsatellite stable colorectal liver metastases and failure with second-line or above therapy, and no subsequent standard treatment regimen.
2. Patients with an ECOG score of 0 or 1, and an expected survival period of ≥6 months.
3. During the study, they are willing to follow the arrangement and not use other systemic anti-tumor drugs such as chemotherapy, targeted, Chinese herbal medicine, and proprietary Chinese medicine.
4. 18-70 years old, no gender limit.

Exclusion Criteria:

1. Those with a history of severe immediate allergy to the drugs used in this study.
2. Cancer patients who require urgent surgical intervention, such as high-risk pathological fractures, life-threatening bleeding symptoms, etc.
3. Any of the following conditions in the 6 months before screening: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient cerebral ischemia Onset or symptomatic pulmonary embolism. Patients with known coronary artery disease, congestive heart failure that does not meet the above criteria or left ventricular ejection fraction <50% must adopt an optimized and stable medical plan determined by the treating doctor. If appropriate, you can consult a cardiologist.
4. Patients with active infection requiring systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1,3,6, and 12 months after completion of radiotherapy
  The proportion of patients showing complete or partial response of low-dose radiotherapy lesions and other metastatic lesions assessed by RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  From the start of treatment to the date of progression or death
Overall survival (OS) | 12 months
  the time from the start of treatment to death from any cause

OTHER OUTCOMES:
Safety evaluation | 12 months
  NCI-CTCAE version 5.0 to assess adverse events (therapeutic toxicity)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China